CLINICAL TRIAL: NCT04023422
Title: Clinic Navigation and Home Visits to Improve Guideline-based Care and Outcomes in Low Income Minority Adults With Asthma
Acronym: HAP3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Andrea Apter, Prinicipal Investigator, Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01HL143364 (NIH)
Record Dates: First submitted 2019-07-12; First posted 2019-07-17 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — House Calls

STUDY DESIGN:
Intervention Model Description: All patients will receive the clinical intervention (CI). In a 2-factor, 2-level factorial design, patients will be randomized to one of four groups by home visitor (HV) and/or physician feedback(CF) intervention: CI + HV, CI + CF, CI + HV + CF, CI. Well-suited for the investigation of the separate components of an intervention, a factorial design permits simple and powerful comparisons between the two factors (home visitor (HV) and clinician feedback CF), cell specific contrasts (the addition of home visitors among patients who have no physician feedback), and the interaction of both interventions. Each patient will be followed over time, so that the additional power of the factorial design will complement the confounder control inherent in randomization plus longitudinal analysis.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Clinical intervention (Active Comparator): Clinical health navigator, a community health worker, facilitates preparation for, attends, and confirms patients's understanding of an office visit.
  Interventions: Behavioral: Clinical intervention; Behavioral: Feedback
- Clinical intervention AND Home Visit (Experimental): Patient receives Clinical intervention and Home visits. Care coordination activities occur taking into account the home environment, its social and physical characteristics.
  Interventions: Behavioral: Clinical intervention; Behavioral: Feedback
- Clinical intervention AND Feedback (Experimental)
  Interventions: Behavioral: Clinical intervention; Behavioral: Feedback
- Clinical intervention AND Home Visit AND Feedback (Experimental)
  Interventions: Behavioral: Clinical intervention; Behavioral: Feedback

INTERVENTIONS:
Behavioral: Clinical intervention — The community health navigator will ask patient to produce medications, to indicate if there are current smokers in the home, to look for structural problems within the home, presence of pests, allergens, pollutants. Pt will be asked to produce their current medications. At the end a report will be written for the clinician.
  Other Names: Home Visit
Behavioral: Feedback — The community health navigator will give the clinician real-time feedback on guideline-related health.

SUMMARY:
Asthma-related deaths are more numerous among low-income minority patients and older adults with chronic diseases. Guidelines for asthma management have not addressed the needs of these groups. The investigators recently demonstrated the feasibility, acceptability, and evidence of effectiveness of two interventions to improve access to care, patient-provider communication, and asthma outcomes: 1) CI: clinic intervention using a patient advocate to prepare for, attend, and confirm understanding of an office visit, and 2) HV: home visits for care coordination and informing clinicians of home barriers to managing asthma is associated with subsequent improvement in asthma outcomes. This project explores whether these interventions can be combined for greater effectiveness, delivery of guideline-based asthma care, and outcomes in low-income minority patients.

In a randomized controlled factorial trial, 400 adults with uncontrolled asthma living in low-income urban neighborhoods are offered 18-months' participation: 12 months of clinical intervention and 6 months of evaluation to monitor sustainability of interventions and outcomes. Patients will be randomized to 1) a patient advocate and (2) an advocate and home visits, (3) an advocate and real-time feedback to the asthma provider (clinician) at each clinic visit of guidelines-relevant relevant information, and 4) (2), and (3). Interventions will be delivered by a community health worker. The study estimates Specific Aim 1: improvement over time of within-group (before-after in four groups) asthma outcomes (asthma control, quality of life, ED visits, hospitalizations, prednisone bursts) Specific Aim 2: across group differences in improvement over time in asthma outcomes; Specific Aim 3: the costs associated with each of the interventions. A cost-offset analysis will determine which intervention costs are offset by savings attributable to reductions in ED, hospitalization or other visits for asthma control and other outcomes.

Exploratory Aim: changes in behavior from the interventions using interviews of clinicians and patients.

Investigators hypothesize that improved outcomes in asthma patients will result from enhanced patient-clinician communication, clinician attention to home environmental exposures, and clinician consideration of the guidelines, at a program cost offset by lower patient health care utilization.

DETAILED DESCRIPTION:
Asthma, a chronic but treatable disease, affects 18.7 million US adults. Asthma-related deaths, hospitalizations, and ED visits are more prevalent in low-income and minority patients, especially African Americans and particularly among older adults, many with co-morbidities.

The Expert Panel Report 3 (EPR3) Guidelines for Asthma Diagnosis and Management, currently undergoing revision, is primarily directed at children and young adults. It overlooks older patients, many with comorbidities and many who live in poverty. Action plans are infrequently used and their benefits, strongly recommended by guidelines, have not been evaluated in older or low-income minority adults. Regular use of inhaled steroids, endorsed by the Guidelines for all but the mildest asthma is limited by social and economic barriers, e.g. cost and accessibility of medication. Failure of guidelines to address the barriers of poverty, limited education, poor housing and communication infrastructure, and suboptimal public transportation may promote non-adherence by clinicians.

For these vulnerable adults, the investigators recently demonstrated the feasibility, acceptability, and evidence of effectiveness of two separate interventions to improve access to care, patient-provider communication, and asthma outcomes: 1) a patient advocate (PA) (HAP2 Study (R18 HL116285)) to prepare for, attend, and confirm understanding of an office visit, and 2) community health workers (CHWs) (ARC Study (PCORI AS 1307-05218)) to assess home barriers to asthma management and coordinate care between home and clinic. Both protocols, well-accepted by patients and clinicians, allow prompting, delivery, and testing of guideline recommendations in a tailored real-world setting. Although these studies were designed and initiated separately, patient advocates in the clinic-based study felt that understanding the home circumstances would be beneficial to clinicians making guideline-based recommendations, while the CHWs visiting homes in the second study wanted more communication with treating clinicians. The proposed project combines these interventions by offering all "PA activities", called the Clinic Intervention (CI) and randomizing half to Home Visits (HV). Additionally, in a factorial design half of patients will be randomized to have their clinician receive feedback on guideline-relevant domains recommended for discussion with patients at appointments. The proposed interventions facilitate communication between clinicians and patients, enriched by understanding of the home environment, the unique view of the patient-clinician interaction at appointments, and barriers to asthma management that patients encounter. While the communication focuses on asthma management, it extends to general care coordination of common co-morbidities such as diabetes, hypertension, obesity and patients will be recruited from both primary care and specialty practices. Community Health Navigators (CHNs), who are lay health workers, will deliver the CI in all patients and the HVs in those so randomized. CHNs with close ties to patients' neighborhoods and also embedded in the clinics, will ensure patients' voices are heard in the delivery of guideline-based care and support patients at risk for health disparities, e. g., older adults, those with comorbidities, low income or limited literacy.

In a randomized controlled factorial trial, adults with uncontrolled asthma living in low-income urban neighborhoods will be offered 18-months participation in four groups of 100 each (1) CI only, (2) CI plus Home Visits (HV), (3) CI and clinician feedback, and (4) CI + HV + clinician feedback. Patients will be evaluated quarterly for 12 months and then observed for 6 months to assess sustainability of the intervention. The investigators will estimate:

Specific Aim 1: improvement over time of within-group (before-after in four groups) asthma outcomes (asthma control, quality of life, ED visits, hospitalizations, prednisone bursts) Specific Aim 2: across group differences in improvement over time in asthma outcomes; Specific Aim 3: the costs associated with each of the intervention, and the investigators will conduct a cost-offset analysis to determine which intervention costs are offset by savings attributable to reductions in ED, hospitalizations or other visits for asthma control and other outcomes.

Exploratory Aim: changes in behavior from the interventions using interviews of clinicians and patients.

Hypothesis and Impact: The investigators hypothesize improved outcomes in asthma patients through enhanced communication of patient and clinician, clinician attention to home environmental exposure, and clinician consideration of the guidelines, at a program cost offset by lower patient health care utilization.

ELIGIBILITY:
Inclusion Criteria:

* Female or male > 18 years and living in a Philadelphia neighborhood in which at least 20% of households have incomes below the federal poverty level (19104, 19120, 19121, 19122, 19124, 19125, 19131, 19132, 19133, 19134, 19139, 19140, 19141, 19142, 19143, 19144, 19145, 19146, 19153, 19151)
* A patient in a participating clinic
* Doctor's diagnosis of asthma
* Prescribed an inhaled corticosteroid for asthma
* Required prednisone or an Emergency Department (ED) visit or hospitalization for asthma within 12 months before enrollment.

  * Some patients with a diagnosis of asthma and prescribed inhaled corticosteroid may also have mention of Chronic Obstructive Pulmonary Disease (COPD) in their record, particularly if they smoke. Asthma and COPD are both heterogeneous diseases, and may be impossible to distinguish by clinical characteristics.Both COPD and asthma can have evidence of reversible obstruction and also of irreversible obstruction. It is important not to exclude these patients, sometimes called overlap patients as they may benefit from these interventions.

Exclusion Criteria:

* Severe psychiatric or cognitive problems making it impossible to understand or carry out the protocol;
* Excluded are those with other chronic lung diseases: lung cancer, cystic fibrosis, heart failure, chronic bronchitis, pulmonary hypertension, a candidate or recipient for lung transplant, a history of bronchial thermoplasty.

Excluded are those with more than 20 pack year tobacco use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Asthma Control at baseline | At randomization
  Asthma Control Questionnaire. The questionnaire has a numerical result 0 - 6 based on response to questionnaire, with lower number indicating better control
Asthma Control at 3 months | 3 months
  Asthma Control Questionnaire. The questionnaire has a numerical result 0 - 6 based on response to questionnaire, with lower number indicating better control
Asthma Control at 6 months | 6 months
  Asthma Control Questionnaire. The questionnaire has a numerical result 0 - 6 based on response to questionnaire, with lower number indicating better control
Asthma Control at 9 months | 9 months
  Asthma Control Questionnaire. The questionnaire has a numerical result 0 - 6 based on response to questionnaire, with lower number indicating better control
Asthma Control at 12 months | 12 months
  Asthma Control Questionnaire. The questionnaire has a numerical result 0 - 6 based on response to questionnaire, with lower number indicating better control
Asthma Control at 15 months | 15 months
  Asthma Control Questionnaire. The questionnaire has a numerical result 0 - 6 based on response to questionnaire, with lower number indicating better control
Asthma Control at 18 months | 18 months
  Asthma Control Questionnaire. The questionnaire has a numerical result 0 - 6 based on response to questionnaire, with lower number indicating better control

SECONDARY OUTCOMES:
hospitalizations for asthma | hospitalizations at 3 months
  number of hospitalizations as indicated in the electronic medical record. If no record is available, the patient's report and verified if possible with patients' record from the outside institution will be used
hospitalizations for asthma | hospitalizations at 6 months
  Number of hospitalizations as indicated in the electronic medical record. If no record is available, patient's report and verified if possible with patients' record from the outside institution will be used.
hospitalizations for asthma | hospitalizations at 9 months
  Number of hospitalizations as indicated in the electronic medical record. If no record is available, patient's report and verified if possible with patients' record from the outside institution will be used.
hospitalizations for asthma | hospitalizations at 12 months
  Number of hospitalizations as indicated in the electronic medical record. If no record is available, patient's report and verified if possible with patients' record from the outside institution will be used.
hospitalizations for asthma | hospitalizations at 15 months
  Number of hospitalizations as indicated in the electronic medical record. If no record is available, patient's report and verified if possible with patients' record from the outside institution will be used.
hospitalizations for asthma | hospitalizations at 18 months
  Number of hospitalizations as indicated in the electronic medical record. If no record is available, patient's report and verified if possible with patients' record from the outside institution will be used.patient's report and verified if possible with patients' record from the outside institution
Emergency Department (ED) visits for asthma | 3 months
  Number of ED visits as indicated in the electronic medical record. If no record is available patient's report and verified if possible with patients' record from the outside institution will be used.
Emergency Department (ED) visits for asthma | 6 months
  Number of ED visits as indicated in the electronic medical record. If no record is available patient's report and verified if possible with patients' record from the outside institution will be used.
Emergency Department (ED) visits for asthma | 9 months
  Number of ED visits as indicated in the electronic medical record. If no record is available patient's report and verified if possible with patients' record from the outside institution will be used.
Emergency Department (ED) visits for asthma | 12 months
  Number of ED visits as indicated in the electronic medical record. If no record is available patient's report and verified if possible with patients' record from the outside institution will be used. report and verified if possible with patients' record from the outside institution
Emergency Department (ED) visits for asthma | 15 months
  Number of ED visits as indicated in the electronic medical record. If no record is available patient's report and verified if possible with patients' record from the outside institution will be used.
Emergency Department (ED) visits for asthma | 18 months
  Number of ED visits as indicated in the electronic medical record. If no record is available patient's report and verified if possible with patients' record from the outside institution will be used.
asthma-related quality of life | 3 months
  Score is the mean of the 15-items each scored 1-7. Higher score indicates better quality of life.
asthma-related quality of life | 6 months
  Score is the mean of the 15-items each scored 1-7. Higher score indicates better quality of life.
asthma-related quality of life | 9 months
  Score is the mean of the 15-items each scored 1-7. Higher score indicates better quality of life.
asthma-related quality of life | 12 months
  Score is the mean of the 15-items each scored 1-7. Higher score indicates better quality of life.
asthma-related quality of life | 15 months
  Score is the mean of the 15-items each scored 1-7. Higher score indicates better quality of life.
asthma-related quality of life | 18 months
  Score is the mean of the 15-items each scored 1-7. Higher score indicates better quality of life.
Forced expiratory volume in 1 second (FEV1) | Month 12
  forced vital capacity in 1 second
Forced expiratory volume in 1 second (FEV1) | Month 18
  forced vital capacity in 1 second

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Pennsylvania Health Center, Philadelphia, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania